CLINICAL TRIAL: NCT01322074
Title: The Relation Between Systemic Inflammatory Markers and Acute Pain in TKA
Brief Title: Systemic Inflammation Versus Acute Pain in Total Knee Arthroplasty (TKA)
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Troels Haxholdt Lunn, MD, Hvidovre University Hospital
Other Study IDs: 9991999
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Other Acute Postoperative Pain; Systemic Inflammatory Response Syndrome
Keywords: Acute postoperative pain; systemic inflammation; CRP; IL6
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for C reactive protein and interleukin 6 analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total knee arthroplasty: Patients operated with elective, unilateral total knee arthroplasty.

SUMMARY:
In this study we evaluate if there is a correlation between acute pain and systemic inflammatory markers after total Knee Arthroplasty (TKA).

DETAILED DESCRIPTION:
The correlation between acute pain and systemic inflammatory markers after total Knee Arthroplasty (TKA) is evaluated.

Level of systemic inflammatory markers (CRP and IL6) are measured preoperatively and 4 and 24 hours postoperatively. These measurements are correlated to postoperative pain (a detailed assessment of pain at rest and during ambulation).

We pole blood-samples collected prospectively (from two data set)

ELIGIBILITY:
Inclusion Criteria:

* Elective unilateral primary total knee arthroplasty
* Able to speak and understand danish
* Able to give informed consent

Exclusion Criteria:

* Alcohol or medical abuse
* Allergies to local anesthetics or methylprednisolone
* Age < 18 years old
* Daily use of strong opioids or glucocorticoids
* Pregnancy or breastfeeding (fertile women)
* Bilateral / revision arthroplasty
* Dementia or other cognitive dysfunction
* Diabetic neuropathy, rheumatoid arthritis, and neurologic or psychiatric diseases potentially influencing pain perception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated with total knee arthroplasty
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2009-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Systemic inflammation vs. pain | 1 week
  The correlation between pain and systemic inflammatory markers (CRP and IL6)

CONTACTS AND LOCATIONS:
Locations (1):
- Dep. of Anesthsiology, Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark